CLINICAL TRIAL: NCT02181127
Title: Closed-Loop Glucagon Administration for the Automated Prevention and Treatment of Hypoglycemia
Brief Title: Closed-Loop Glucagon Administration For Hypoglycemia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P001663/MGH
Record Dates: First submitted 2013-09-09; First posted 2014-07-03 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Type 1 Diabetes
Keywords: bionic pancreas; artificial pancreas; insulin; glucagon; continuous glucose monitoring (CGM); outpatient; insulin pump; glucagon pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucagon-only Bionic Pancreas (active) (Active Comparator): Glucagon-only Bionic Pancreas will deliver glucagon during 7 of the 14 days. The order of the glucagon days will be randomized in blocks of 2, with no more than 2 days in a row of glucagon.
  Interventions: Device: Glucagon-only Bionic Pancreas
- Glucagon-only Bionic Pancreas (placebo) (Placebo Comparator): Glucagon-only Bionic Pancreas will deliver placebo during 7 of the 14 days. The order of the placebo days will be randomized in blocks of 2, with no more than 2 days in a row of placebo.
  Interventions: Device: Glucagon-only Bionic Pancreas

INTERVENTIONS:
Device: Glucagon-only Bionic Pancreas — A computer algorithm will automatically deliver glucagon based on the signal from a minimally invasive continuous glucose monitor.
  Other Names: Boston University Bionic Pancreas

SUMMARY:
This study will test the hypothesis that a wearable automated bionic pancreas system that automatically delivers glucagon only can prevent or treat hypoglycemia vs. usual care for people with type 1 diabetes > 21 years old.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older with type 1 diabetes for at least one year.
* Otherwise healthy (mild chronic disease such as asthma, hypertension, and depression will be allowed if well controlled).
* Self-reported frequency of documented hypoglycemia (BG < 60 mg/dl) of at least 2 times per week
* Partial hypoglycemic unawareness (inconsistent symptoms with BG < 50 mg/dl) or hypoglycemic unawareness (minimal or no symptoms with BG < 50 mg/dl)

Exclusion Criteria:

* Unable to provide informed consent.
* Unable to comply with study procedures.
* Current participation in another diabetes-related clinical trial other than one that is primarily observational in nature.
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception
* History of cystic fibrosis, pancreatitis, or other pancreatic disease other than type 1 diabetes
* End stage renal disease on dialysis (hemodialysis or peritoneal dialysis).
* Any known liver or biliary disease including cirrhosis, alcoholic liver disease, non-alcoholic fatty liver disease, non-alcoholic steatohepatitis, any form of viral hepatitis.
* Congestive heart failure (established history of CHF, paroxysmal nocturnal dyspnea, or orthopnea).
* Acute illness or exacerbation of chronic illness at the time of the study.
* Seizure disorder or history of hypoglycemic seizure in the last 1 year
* History of pheochromocytoma. Fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor:
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year).
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days) or substance abuse (any use within the last 6 months of controlled substances without a prescription).
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference.
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
* Unwilling or unable to completely avoid acetaminophen during the study period.
* Any factors that, in the opinion of the principal investigator, would interfere with the safe completion of the study procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about this and related studies — http://bionicpancreas.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 participants were enrolled in the trial, but only 22 participants actually participated. 4 subjects were not eligible to participate. The remaining 5 subjects that did not participate were considered "back up" or "benched" subjects who were eligible and willing to participate, but were not required to meet our desired total cohort.
Groups:
- Glucagon-only Bionic Pancreas: Subjects will use the device every day and will fill the reservoir daily with glucagon or placebo (randomized, double blinded allocation for each day).
  Glucagon-only Bionic Pancreas: A computer algorithm will automatically deliver glucagon based on the signal from a minimally invasive continuous glucose monitor.
Period: Overall Study
Arm/Group | Glucagon-only Bionic Pancreas
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Continuous Glucose Monitor (CGM) Glucose Total Area Over the Curve and Less Than 60 mg/dl
Time Frame: From t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: mg/dl/min
Groups:
- Glucagon-only Bionic Pancreas: Glucagon-only Bionic Pancreas delivered glucagon during 7 of the 14 days. The order of the glucagon days was randomized in blocks of 2, with no more than 2 days in a row of glucagon.
- Placebo: Glucagon-only Bionic Pancreas delivered placebo during 7 of the 14 days. The order of the placebo days was randomized in blocks of 2, with no more than 2 days in a row of placebo.
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
mg/dl/min | 1015 (883.24) | 4375.68 (3058.77)

2. Secondary Outcome: Percentage of Time CGM Glucose Less Than 70 mg/dl Overnight and During Daytime
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 22
percentage of time
  Glucagon - daytime | 3.92 (2.42)
  Glucagon - overnight | 1.50 (2.18)
  Placebo - daytime | 7.94 (4.62)
  Placebo - overnight | 10.25 (7.15)

3. Secondary Outcome: Number of Hypoglycemic Episodes With CGMG < 50 mg/dl
Time Frame: From t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
number of episodes | 1.73 (1.39) | 5.0 (3.07)

4. Secondary Outcome: Number of Hypoglycemic Episodes With CGMG < 60 mg/dl
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
number of episodes | 4.14 (2.23) | 8.86 (4.57)

5. Secondary Outcome: Number of Hypoglycemic Episodes With CGMG < 70 mg/dl
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
number of episodes | 8.95 (5.55) | 12.68 (5.54)

6. Secondary Outcome: Fraction of Time Spent Within Each of the Following Glucose Ranges as Determined From All CGMG Measurements: < 70 mg/dl,70-120 mg/dl,70-180 mg/dl, >180 mg/dl, >250 mg/dl
Time Frame: from t=0 to stud stop after 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
percentage of time
  CGMG < 70 mg/dl | 3.11 (2.02) | 8.73 (5.10)
  CGMG 70-120 mg/dl | 33.32 (15.85) | 30.53 (14.74)
  CGMG 70-180 mg/dl | 68.91 (15.39) | 61.89 (13.79)
  CGMG > 180 mg/dl | 27.98 (16.44) | 29.38 (15.74)
  CGMG > 250 mg/dl | 9.05 (8.05) | 9.83 (8.14)

7. Secondary Outcome: Count of Subjects With Mean CGMG < 154mg/dl
Time Frame: from t=0 to study stop after 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 13 | 11

8. Secondary Outcome: Mean CGMG During Exercise
Description: Times of exercise were not collected during the study, and therefore this outcome cannot be calculated.
Time Frame: 2 weeks
Population: Times of exercise were not collected during the study, and therefore this outcome cannot be calculated.
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

9. Secondary Outcome: Mean Absolute Relative Deviation (MARD) vs. Subset of BG Measurements Before Meals and at Bedtime
Description: Blood sugar measurements were not specified as before meals and before bed during the study, so we are unable to calculate and report this outcome.
Time Frame: 2 weeks
Population: Blood sugar measurements were not specified as before meals and before bed during the study, so we are unable to calculate and report this outcome.
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

10. Secondary Outcome: Mean Absolute Relative Deviation (MARD) Between Capillary Blood Glucose and CGM Glucose Values
Description: Paired values between the blood glucose measurements and CGM glucose measurements were compared, and the percent difference was recorded. The mean of the absolute value of all the differences is reported here, and reflects the accuracy of the CGM glucose measurements relative to the capillary blood glucose measurements.
Time Frame: from t=0 to study stop after 2 weeks
Population: This analysis is not broken down according to randomization, because it is intended to give context to the other CGM reported outcomes by reflecting the accuracy of the CGM.
Measure: Mean (Standard Deviation); unit: percent difference
Groups:
- All Participants: All participants in the study, on both glucagon and placebo days
Arm/Group | All Participants
Number analyzed (Participants) | 22
percent difference | 15.20 (14.56)

11. Secondary Outcome: Number of Hypoglycemic Events (< 60 mg/dl) as Determined From BG Measurements
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
number of events | 0.73 (0.98) | 2.59 (2.59)

12. Secondary Outcome: Average BG as Determined From the Measurements Taken Before Meals and Before Bedtime
Description: as for outcome 9
Time Frame: 2 weeks
Population: as for outcome 9
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of the BG Values Taken Before Meals and Before Bedimte Less Than 70 mg/dl
Description: as for outcome 9
Time Frame: 2 weeks
Population: as for outcome 9
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of All BG Values Less Than 70 mg/dl
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: number of values
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
number of values | 1.45 (1.99) | 4.23 (3.90)

15. Secondary Outcome: Number of Study Days With Mean BG < 154 mg/dl
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
number of days | 4.4 (2.2) | 4.2 (2.2)

16. Secondary Outcome: Fraction Measurements Within Each of the Following Glucose Ranges as Determined From HemoCue Measurements Taken Before Meals and Before Bed: < 70 mg/dl,70-120 mg/dl,70-180 mg/dl,>180 mg/dl,>250 mg/dl
Description: as for outcome 9
Time Frame: 2 weeks
Population: as for outcome 9
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

17. Secondary Outcome: Mean BG During Exercise
Description: Times of exercise were not collected during the study, and therefore this outcome cannot be calculated.
Time Frame: 2 weeks
Population: Times of exercise were not collected during the study, and therefore this outcome cannot be calculated.
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

18. Secondary Outcome: • Fraction of BG Values < 70 During Exercise Fraction of BG Values < 70 During Exercise
Description: Times of exercise were not collected during the study, and therefore this outcome cannot be calculated.
Time Frame: 2 weeks
Population: Times of exercise were not collected during the study, and therefore this outcome cannot be calculated.
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

19. Secondary Outcome: Number of Carbohydrate Interventions for Hypoglycemia
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: number of interventions per day
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
number of interventions per day | 1.25 (0.48) | 1.89 (0.83)

20. Secondary Outcome: Total Number of Grams of Carbohydrate Taken for Hypoglycemia
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
grams per day | 23.90 (9.52) | 36.29 (22.95)

21. Secondary Outcome: Insulin Total Daily Dose
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: units per day
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
units per day | 38.7 (12.6) | 37.0 (12.0)

22. Secondary Outcome: • Number of Carbohydrate Interventions for Hypoglycemia During the Daytime (7:00 AM - 11:00 PM)
Description: Timing of carbohydrate consumption for treatment of hypoglycemia was not collected during the study, so this outcome cannot be calculated
Time Frame: 2 weeks
Population: Timing of carbohydrate consumption for treatment of hypoglycemia was not collected during the study, so this outcome cannot be calculated
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

23. Secondary Outcome: Total Number of Grams of Carbohydrate Taken for Hypoglycemia During the Daytime (7:00 AM - 11:00 PM)
Description: as for outcome 22
Time Frame: 2 weeks
Population: as for outcome 22
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

24. Secondary Outcome: Number of Carbohydrate Interventions for Hypoglycemia Overnight (11:00 PM - 7:00 AM)
Description: as for outcome 22
Time Frame: 2 weeks
Population: as for outcome 22
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

25. Secondary Outcome: Total Number of Grams of Carbohydrate Taken for Hypoglycemia Overnight (11:00 PM - 7:00 AM)
Description: as for outcome 22
Time Frame: 2 weeks
Population: as for outcome 22
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 0

26. Secondary Outcome: Total Glucagon Dosing (mcg/kg/24 Hours)
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: mcg/kg/day
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
mcg/kg/day | 6.84 (2.90) | 9.8 (3.6)

27. Secondary Outcome: Episodes of Nausea Per Day on Glucagon vs Placebo
Time Frame: from t=0 to study stop after 2 weeks
Measure: Mean (Standard Deviation); unit: episodes of nausea per day
Arm/Group | Glucagon-only Bionic Pancreas | Placebo
Number analyzed (Participants) | 22 | 22
episodes of nausea per day | 1.1 (1.6) | 0.4 (.07)

ADVERSE EVENTS:
Arm/Group | Glucagon-only Bionic Pancreas
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No